CLINICAL TRIAL: NCT02275338
Title: An International, Multicentric, Prospective, Open Label Study to Assess the Efficacy and Safety of Lanreotide Autogel 120 MG Associated to Standard of Care in the Treatment of Clinical Symptoms Associated With Inoperable Malignant Intestinal Obstruction
Brief Title: Study to Assess Efficacy and Safety of Lanreotide Autogel 120 MG in Treatment of Clinical Symptoms Associated With Inoperable Malignant Intestinal Obstruction
Acronym: IMIO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: A-48-52030-269; 2013-002174-43 (EudraCT Number)
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Intestinal Obstruction
MeSH Terms: conditions — Intestinal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lanreotide Autogel (Experimental): 120mg administered via deep subcutaneous injection at Day 0 and Day 28.
  Interventions: Drug: Lanreotide Autogel

INTERVENTIONS:
Drug: Lanreotide Autogel — 120mg administered via deep subcutaneous injection at Day 0 and Day 28.
  Other Names: Somatuline Autogel

SUMMARY:
To assess the efficacy of Lanreotide Autogel 120 mg for the relief of vomiting due to inoperable malignant intestinal obstruction in patients without nasogastric tube (NGT) and to assess the efficacy of lanreotide Autogel 120 mg on removal of nasogastric tube without the recurrence of vomiting in patients with an inoperable malignant intestinal obstruction with a nasogastric tube.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before any study related procedure
* Male and female patients age 18 years or older at time of enrollment
* Diagnosis of intestinal obstruction of malignant origin
* In case of peritoneal carcinomatosis, confirmation by CT or MRI scan within the 3 months preceding the inclusion in the study
* Confirmed as inoperable after surgical advice
* Patient with a nasogastric tube OR presenting with 3 or more episodes of vomiting / 24h in the last 48 hours
* Estimated life expectancy 1 month or more

Exclusion Criteria:

* Operable obstruction or subobstruction
* Bowel obstruction due to a non-malignant cause
* Signs of bowel perforation
* Prior treatment with somatostatin or any other analogue within the previous 60 days
* A known hypersensitivity to any of the study treatments or related compounds
* Previous participation in this study
* Is likely to require treatment during the study with drugs that are not permitted by the study protocol
* Has abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardise the subject's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (17):
- Belgium (17):
  - Aalst
  - Antwerp
  - Bruges
  - Ste-Elisabeth Hospital, Brussels
  - Chimay
  - Ghent
  - Haine-Saint-Paul
  - Libramont
  - Liège
  - Mons
  - Montigny-le-Tilleul
  - Ostend
  - Ottignies
  - Sint-Niklaas
  - Tournai
  - Verviers
  - Yvoir

REFERENCES:
- [Derived] Duck L, Demolin G, D'Hondt L, Dopchie C, Hendrickx K, Lannoye B, Bastin F, Lossignol D, Hamdan O, Lybaert W, Vandenhaute V, Regnault B, De Ruyter V, Geboes K. Efficacy and Safety of Lanreotide Autogel in the Treatment of Clinical Symptoms Associated With Inoperable Malignant Intestinal Obstruction: A Prospective Phase II Study. Clin Ther. 2021 Dec;43(12):2136-2145.e2. doi: 10.1016/j.clinthera.2021.10.014. Epub 2021 Nov 26. PMID 34844770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects diagnosed with inoperable malignant intestinal obstruction were recruited into this single arm, open label study in 15 study centres in Belgium between November 2014 and November 2017.
Pre-assignment Details: Overall, 52 subjects were enrolled into this 2 phase study.
Groups:
- Lanreotide Autogel® 120 mg - All Subjects: All subjects were administered an initial injection of lanreotide Autogel® 120 milligrams (mg) via subcutaneous injection at Day 0 (Phase 1).
  Subjects who completed the 28 days of Phase 1 and who were responders as defined by the protocol, had the opportunity to enter Phase 2 and receive a second subcutaneous injection of lanreotide Autogel® 120 mg.
  All subjects continued to receive standard of care throughout the study.
Period: Overall Study
Arm/Group | Lanreotide Autogel® 120 mg - All Subjects
Started | 52
Completed Phase 1 | 25
Started Phase 2 | 21
Completed | 19
Not Completed | 33
Not completed — Adverse Event | 15
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 4
Not completed — Disease progression (death) | 1
Not completed — Ineligible to start Phase 2 | 4
Not completed — Reason not specified | 5
Not completed — Does not meet entry criteria | 1

BASELINE CHARACTERISTICS:
Population: All subjects who received at least 1 dose of study medication (Intention to Treat [ITT] population).
Groups:
- Lanreotide Autogel® 120 mg - All Subjects: All subjects were administered an initial injection of lanreotide Autogel® 120 mg via subcutaneous injection at Day 0 (Phase 1).
  Subjects who completed the 28 days of Phase 1 and who were responders as defined by the protocol, had the opportunity to enter Phase 2 and receive a second subcutaneous injection of lanreotide Autogel® 120 mg.
  All subjects continued to receive standard of care throughout the study.
Arm/Group | Lanreotide Autogel® 120 mg - All Subjects
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (12.1)
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 1
  40-49 years | 3
  50-59 years | 9
  60-69 years | 17
  >= 70 years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 51
  More than one race | 0
  Unknown or Not Reported | 0
Nasogastric tube (NGT) Status at Baseline [Count of Participants; unit: Participants]
  With NGT at baseline | 35
  Without NGT at baseline | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders Before or at Day 7
Description: The primary endpoint assessed the percentage of responding subjects before or at Day 7. A responder was defined as a subject experiencing ≤2 vomiting episodes/day during at least 3 consecutive days at any timepoint between Day 0 and Day 7 (for subjects without NGT at baseline), or as a subject in whom the NGT had been removed during at least 3 consecutive days at any timepoint between Day 0 and Day 7 without vomiting recurrence (for subjects with NGT at baseline), as recorded on diary cards which were completed every day.
Time Frame: From Day 0 to Day 7
Population: All subjects who received at least 1 dose of study medication (ITT population).
Measure: Number; unit: percentage of responders
Groups:
- Lanreotide Autogel® 120 mg: All subjects were administered an initial injection of lanreotide Autogel® 120 mg via subcutaneous injection at Day 0 (Phase 1).
  Subjects who completed the 28 days of Phase 1 and who were responders as defined by the protocol, had the opportunity to enter Phase 2 and receive a second subcutaneous injection of lanreotide Autogel® 120 mg.
  All subjects continued to receive standard of care throughout the study.
Arm/Group | Lanreotide Autogel® 120 mg
Number analyzed (Participants) | 52
percentage of responders
  Without NGT at Baseline: number analyzed (Participants) | 17
  Without NGT at Baseline | 88.2
  With NGT at Baseline: number analyzed (Participants) | 35
  With NGT at Baseline | 25.7
  All Subjects | 46.2
Statistical Analysis 1: Comparison: Lanreotide Autogel® 120 mg; One sided binomial test to compare percentage of responding subjects to theoretical proportion of 30%; Test type: Other; p = 0.0055, Binomial test — The expected proportion of responders using Lanreotide was 50%, 1 sided test, 2.5% significance level alpha and power of 80% using Z-test for binomial proportion

2. Secondary Outcome: Percentage of Responders in Phase 1
Description: This endpoint assessed the overall percentage of responding subjects at the Phase 1 timepoints of Days 14 and 28. A responder was defined as a subject experiencing ≤ 2 vomiting episodes/day during at least 3 consecutive days at any timepoint between Day 0 and Days 14 or 28 (for subjects without NGT at baseline) or as a subject in whom the NGT has been removed, during at least 3 consecutive days without vomiting recurrence, at any timepoint between Day 0 and Days 14 and 28 (for subjects with NGT at baseline), as recorded on diary cards which were completed every day.
Time Frame: From Day 0 to Day 28
Population: All subjects who received at least 1 dose of study medication (ITT population).
Measure: Number; unit: percentage of responders
Arm/Group | Lanreotide Autogel® 120 mg - All Subjects
Number analyzed (Participants) | 52
percentage of responders
  By Day 14: Without NGT at Baseline: number analyzed (Participants) | 17
  By Day 14: Without NGT at Baseline | 88.2
  By Day 14: With NGT at Baseline: number analyzed (Participants) | 35
  By Day 14: With NGT at Baseline | 45.7
  By Day 14: All Subjects | 59.6
  By Day 28: Without NGT at Baseline: number analyzed (Participants) | 17
  By Day 28: Without NGT at Baseline | 88.2
  By Day 28: With NGT at Baseline: number analyzed (Participants) | 35
  By Day 28: With NGT at Baseline | 54.3
  By Day 28: All Subjects | 65.4

3. Secondary Outcome: Median Time Between First Lanreotide Autogel® Injection and Clinical Response in Phase 1
Description: The time for clinical response in Phase 1 (up to Day 28) was defined as the time from inclusion (Day 0) to the date of clinical response. A response was defined as occurrence of ≤ 2 vomiting episodes/day for at least 3 consecutive days at any timepoint between Day 0 and Day 28 (for patients without NGT use at baseline) or the removal of NGT for at least 3 consecutive days at any timepoint between Day 0 and Day 28 without vomiting recurrence (for patients with NGT use at baseline). The Kaplan-Meier estimate of median time to clinical response are presented.
Time Frame: From Day 0 to Day 28
Population: All subjects who received at least 1 dose of study medication (ITT population).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lanreotide Autogel® 120 mg - All Subjects
Number analyzed (Participants) | 52
days | 9.00 [5.00 to 14.00]

4. Secondary Outcome: Median Change From Baseline in Quality of Life as Assessed by Edmonton Symptom Assessment System (ESAS) in Phase 1
Description: Quality of Life was assessed by both subject and investigator based on the ESAS. The ESAS scale evaluates 9 symptoms common in cancer subjects: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing and shortness of breath. The severity at the time of assessment of each symptom is rated from 0 to 10 on a numerical scale; 0 = symptom is absent and 10 = worst possible severity. Each symptom rating was interpreted independently and a total symptom distress score was calculated for both subject and investigator assessed scores as the sum of the 9 items. Median change from baseline (Day 0) in total symptom distress score, at each of the Phase 1 timepoints is presented and a positive change indicates a worsening condition.
Time Frame: Days 0, 7, 14 and 28
Population: All subjects who received at least 1 dose of study medication (ITT population). Only subjects with data available for analysis at each timepoint are presented.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lanreotide Autogel® 120 mg - All Subjects
Number analyzed (Participants) | 52
units on a scale
  Day 7 - assessed by subject: number analyzed (Participants) | 33
  Day 7 - assessed by subject | -3.0 [-11.0 to 1.0]
  Day 7 - assessed by investigator: number analyzed (Participants) | 28
  Day 7 - assessed by investigator | -4.5 [-14.0 to 3.0]
  Day 14 - assessed by subject: number analyzed (Participants) | 34
  Day 14 - assessed by subject | -2.0 [-14.0 to 1.0]
  Day 14 - assessed by investigator: number analyzed (Participants) | 28
  Day 14 - assessed by investigator | -7.5 [-17.0 to 2.0]
  Day 28 - assessed by subject: number analyzed (Participants) | 18
  Day 28 - assessed by subject | -5.5 [-14.0 to -1.0]
  Day 28 - assessed by investigator: number analyzed (Participants) | 20
  Day 28 - assessed by investigator | -5.0 [-14.0 to 5.5]

5. Secondary Outcome: Median Change From Baseline in General Activity as Assessed by the Karnofsky Performance Status (KPS) Scale in Phase 1
Description: The KPS scale was used to quantify subject's general well-being and activities of daily life. Subjects were classified based on their functional impairment and KPS scores range from 0 (death) to 100 (no evidence of disease). KPS scores are classified as 0-40 = unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly; 50-70 = unable to work; able to live at home and care for most personal needs; varying amount of assistance needed; 80-100 = able to carry on normal activity and to work; no special care needed. Median change from baseline (Day 0) at each of the Phase 1 timepoints is presented and a negative change indicates a worsening condition.
Time Frame: Days 0, 7, 14 and 28
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lanreotide Autogel® 120 mg - All Subjects
Number analyzed (Participants) | 52
units on a scale
  At Day 7: number analyzed (Participants) | 41
  At Day 7 | 0.0 [0.0 to 10.0]
  At Day 14: number analyzed (Participants) | 36
  At Day 14 | 0.0 [0.0 to 20.0]
  At Day 28: number analyzed (Participants) | 25
  At Day 28 | 10.0 [0.0 to 30.0]

6. Secondary Outcome: Median Change From Baseline in Number of Daily Episodes of Nausea in Phase 1
Description: The mean number of daily episodes of nausea were calculated as the sum of episodes of nausea reported the last 3 days before the corresponding visit, divided by 3.
  The median change from baseline (Day 0) at each of the Phase 1 timepoints is presented and positive change indicates a worsening condition.
Time Frame: Days 0, 7, 14 and 28
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Daily episodes of nausea
Arm/Group | Lanreotide Autogel® 120 mg - All Subjects
Number analyzed (Participants) | 52
Daily episodes of nausea
  At Day 7: number analyzed (Participants) | 16
  At Day 7 | -0.17 [-1.67 to 0.0]
  At Day 14: number analyzed (Participants) | 14
  At Day 14 | -1.50 [-4.00 to 0.00]
  At Day 28: number analyzed (Participants) | 12
  At Day 28 | -1.50 [-3.67 to 0.00]

7. Secondary Outcome: Median Change From Baseline in Abdominal Pain Scores Assessed Using Visual Analogue Scale (VAS) in Phase 1
Description: Abdominal pain was assessed using the VAS numeric pain distress scale. The VAS is a 100-millimetre (10-centimetre) scoring scale on which subjects marked on their perceived level of pain. Score range on VAS is from 0 to 100 where 0 = no pain and 100 = unbearable pain. Median change from baseline (Day 0) at each of the Phase 1 timepoints is presented and a positive change indicates a worsening condition.
Time Frame: Days 0, 7, 14 and 28
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lanreotide Autogel® 120 mg - All Subjects
Number analyzed (Participants) | 52
units on a scale
  At Day 7: number analyzed (Participants) | 39
  At Day 7 | -3.0 [-13.0 to 0.0]
  At Day 14: number analyzed (Participants) | 37
  At Day 14 | -1.0 [-9.0 to 6.0]
  At Day 28: number analyzed (Participants) | 23
  At Day 28 | 0.0 [-9.0 to 10.0]

8. Secondary Outcome: Percentage of Responders Before or at Phase 2 Timepoints
Description: This endpoint assessed the overall percentage of subjects continuing from Phase 1 and confirmed as a responder at the end of Phase 1, showing a continued response at Days 35, 42 and 56. A responder was defined as a subject experiencing ≤2 vomiting episodes/day during at least 3 consecutive days at any timepoint between Day 0 and Days 35, 42, 56 (for subjects without NGT at baseline), or as a subject in whom the NGT had been removed during at least 3 consecutive days at any timepoint between Day 0 and Days 35, 42, 56 without vomiting recurrence (for subjects with NGT at baseline), as recorded on diary cards which were completed every day.
Time Frame: From Day 0 to Day 56
Population: All subjects who received at least 1 dose of study medication (ITT population) and were continuing in Phase 2 of the study.
Measure: Number; unit: percentage of responders
Arm/Group | Lanreotide Autogel® 120 mg - All Subjects
Number analyzed (Participants) | 21
percentage of responders
  By Day 35: Without NGT at Baseline: number analyzed (Participants) | 10
  By Day 35: Without NGT at Baseline | 100
  By Day 35: With NGT at Baseline: number analyzed (Participants) | 11
  By Day 35: With NGT at Baseline | 100
  By Day 35: All Subjects | 100
  By Day 42: Without NGT at Baseline: number analyzed (Participants) | 10
  By Day 42: Without NGT at Baseline | 100
  By Day 42: With NGT at Baseline: number analyzed (Participants) | 11
  By Day 42: With NGT at Baseline | 100
  By Day 42: All Subjects | 100
  By Day 56: Without NGT at Baseline: number analyzed (Participants) | 10
  By Day 56: Without NGT at Baseline | 100
  By Day 56: With NGT at Baseline: number analyzed (Participants) | 11
  By Day 56: With NGT at Baseline | 100
  By Day 56: All Subjects (n=21) | 100

9. Secondary Outcome: Median Change From Baseline in Quality of Life as Assessed by ESAS in Phase 2
Description: Quality of Life was assessed by both subject and investigator based on the ESAS. The ESAS scale evaluates 9 symptoms common in cancer subjects: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing and shortness of breath. The severity at the time of assessment of each symptom is rated from 0 to 10 on a numerical scale, 0 = symptom is absent and 10 = worst possible severity. Each symptom rating was interpreted independently and a total symptom distress score was calculated for both subject and investigator assessed scores as the sum of the 9 items. Median change from baseline (Day 0) in total symptom distress score, at each of the Phase 2 timepoints is presented and a positive change indicates a worsening condition.
Time Frame: Days 0, 35, 42 and 56
Population: All subjects who received at least 1 dose of study medication (ITT population) and were continuing in Phase 2 of the study. Only subjects with data available for analysis at each timepoint are presented.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lanreotide Autogel® 120 mg - All Subjects
Number analyzed (Participants) | 21
units on a scale
  Day 35 - assessed by subject: number analyzed (Participants) | 18
  Day 35 - assessed by subject | -4.0 [-22.0 to 1.0]
  Day 35 - assessed by investigator: number analyzed (Participants) | 18
  Day 35 - assessed by investigator | -12.0 [-18.0 to -2.0]
  Day 42 - assessed by subject: number analyzed (Participants) | 16
  Day 42 - assessed by subject | -10.5 [-16.0 to 0.0]
  Day 42 - assessed by investigator: number analyzed (Participants) | 14
  Day 42 - assessed by investigator | -13.5 [-19.0 to -3.0]
  Day 56 - assessed by subject: number analyzed (Participants) | 17
  Day 56 - assessed by subject | -8.0 [-17.0 to -1.0]
  Day 56 - assessed by investigator: number analyzed (Participants) | 17
  Day 56 - assessed by investigator | -9.0 [-17.0 to -2.0]

ADVERSE EVENTS:
Time Frame: All cause mortality and Adverse events (AEs) were monitored from the time the subject gave informed consent (Day 0) and throughout the study up to Day 56.
Description: The safety analysis population includes all subjects who received at least 1 dose of study medication.
Arm/Group | Lanreotide Autogel® 120 mg - All Subjects
All-Cause Mortality (participants affected / at risk) | 15/52
Serious Adverse Events (participants affected / at risk) | 29/52
Other Adverse Events (participants affected / at risk) | 38/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel® 120 mg - All Subjects (N=52)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Disease progression (General disorders) | 9 (9)
General physical health deterioration (General disorders) | 3 (3)
Inflammation (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Abscess intestinal (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Paresis (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Explorative laparotomy (Surgical and medical procedures) | 1 (1)
Small intestinal resection (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel® 120 mg - All Subjects (N=52)
Anaemia (Blood and lymphatic system disorders) | 10 (24)
Neutropenia (Blood and lymphatic system disorders) | 5 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (8)
Abdominal pain (Gastrointestinal disorders) | 9 (11)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 10 (12)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 9 (10)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Asthenia (General disorders) | 5 (5)
Fatigue (General disorders) | 6 (6)
Inflammation (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (5)
Pollakiuria (Renal and urinary disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypertension (Vascular disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 10 (13)

LIMITATIONS AND CAVEATS:
Results from outcome measures regarding change from baseline in quality of life (ESAS scale), general activity (KPS Scale) and daily episodes of nausea should be interpreted with caution due to small sample sizes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-10-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT02275338/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT02275338/SAP_001.pdf